CLINICAL TRIAL: NCT04083014
Title: An Open, One-arm, Prospective Study of a Single Dose Anti-CD20 Monoclonal Antibody Combined With Bortezomib for Treatment of Relapsed Refractory Autoimmune Hemolytic Anemia
Brief Title: Single-dose Anti-CD20 Antibody With Bortezomib for Relapsed Refractory Autoimmune Hemolytic Anemia
Acronym: RRAIHA01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Chen Miao, associate professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2053
Record Dates: First submitted 2019-08-31; First posted 2019-09-10 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Autoimmune Hemolytic Anemia; Autoimmune Hemolytic Anemia and Autoimmune Thrombocytopenia
Keywords: warm autoimmune hemolytic anemia; relapsed; refractory; EVANS syndrome; anti-CD20 monoclonal antibody; bortezomib
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Evans Syndrome; Recurrence | interventions — Bortezomib; Rituximab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): The treatment regimen is a single dose anti-CD20 antibody injection (500mg iv drip，day0) combined with bortezomib injection (1.3mg/m2 subcutaneous injection，twice a week for two weeks，day1，4，8，11). The treatment course will be repeated three months later.
  Interventions: Drug: combination of a single dose anti-CD20 antibody and bortezomib

INTERVENTIONS:
Drug: combination of a single dose anti-CD20 antibody and bortezomib — Relapsed and refractory warm AIHA patients receive treatment of combination of a single dose anti-CD20 antibody and bortezomib twice during three months interval.
  Other Names: Rituximab Injection; Bortezomib for Injection

SUMMARY:
Patients of relapsed and refractory warm autoimmune hemolytic anemia or EVANS syndrome aged 18 to 80 will be included in this study. The treatment regimen is a single dose anti-CD20 antibody (500mg) combined with bortezomib (1.3mg/m2 twice a week for two weeks). The treatment course would be repeated three months later.

DETAILED DESCRIPTION:
Glucocorticoids are the first-line treatment of warm AIHA. The overall response is 70-90%, but 10% to 20% patients are refractory to GCs and more than 50% patients will relapse after GCs tapering or cessation.

Anti-CD20 monoclonal antibody is the preferred second-line treatment for relapsed refractory wAIHA. Anti-CD20 antibody 375 mg/m2, once a week, four times, is the standard treatment regimen. Low dose anti-CD20 antibody, 100mg once a week, four times, also showed similar response rate. However, the use of four times of intravenous infusion is trouble. So the investigators intend to explore the efficiency of the singe dose of 500mg anti-CD20 antibody.

Anti-CD20 antibody takes median 6-8 weeks to response and only about 50% patients achieving long-term response. Plasma cells produce antibodies and long-lived plasma cells in bone marrow and spleen continuously work. Bortezomib is a proteasome inhibitor and targets plasma cells. Bortezomib has become a first-line treatment for clonal plasma cell diseases (such as multiple myeloma, systemic amyloidosis, POEMS syndrome, etc.). Bortezomib can also induce reactive plasma cell apoptosis and has a variety of immunomodulatory effects. The investigators try to combine bortezomib with anti-CD20 antibody, which may play a synergistic role and improve the efficacy.

Patients of relapsed and refractory warm autoimmune hemolytic anemia or EVANS syndrome will receive a single dose anti-CD20 antibody (500mg) and bortezomib (1.3mg/m2 twice a week for two weeks) twice for three months interval.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of warm autoimmune hemolytic anemia or EVANS syndrome, primary or secondary.
2. Patients refractory to glucocorticoids (HGB increase less than 20g/L after three weeks full dose glucocorticoids treatment). Or patients relapse after at least one course of glucocorticoids therapy (HGB < 110g/L in female and HGB < 120g/L in male). Or glucocorticoids dependence (prednisone maintenance dose > 10mg a day). Or glucocorticoids intolerance.
3. Normal heart function, liver function (total bilirubin < 1.5×ULN, ALT, AST < 3.0 ×ULN), and renal function (serum creatinine < 1.0 ×ULN).
4. No active infection.
5. No malignant tumors (except carcinoma in situ).
6. Patients understand the content of the study, participate the study and sign the informed consent voluntarily.

Exclusion Criteria:

1. Patients with malignant tumors (excluding carcinoma in situ);
2. With uncontrollable infections or other serious diseases;
3. Active hepatitis B, serume HBV-DNA > 104copies/ml;
4. Women during pregnancy or lactation;
5. Not strict contraception;
6. Psychiatric patients and those with severe mental illness.
7. Other conditions that researchers consider inappropriate to join the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
response time | two years
  days hemoglobin increasing more than 20g/L
overall response | two years
  total of complete response and partial response
complete response | two years
  rate of achieving complete response
relapse rate | two years
  relapse rate of responders

SECONDARY OUTCOMES:
relapse free survival | two years
  time duration of responders from first treatment to recurrence of decompensated hemolysis
overall survival | two years
  time from first treatment to death of any causes
side effects | two years
  side effects due to the combination of anti-CD20 antibody and bortezomib

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Patients age,gender,diagnosis,treatment details, efficiency and survival.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available 6 months after the publication of the study and for 2 years.
Access Criteria: get permission from the researchers.

REFERENCES:
- [Background] Lechner K, Jager U. How I treat autoimmune hemolytic anemias in adults. Blood. 2010 Sep 16;116(11):1831-8. doi: 10.1182/blood-2010-03-259325. Epub 2010 Jun 14. PMID 20548093
- [Background] Group, Chinese Society of Hematology, Chinese Medical Association. [Chinese expert consensus on the diagnosis and treatment of autoimmune hemolytic anemia (2017) Red Blood Cell Disease (Anemia)]. Zhonghua Xue Ye Xue Za Zhi. 2017 Apr 14;38(4):265-267. doi: 10.3760/cma.j.issn.0253-2727.2017.04.001. No abstract available. Chinese. PMID 28468084
- [Background] Hill A, Hill QA. Autoimmune hemolytic anemia. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):382-389. doi: 10.1182/asheducation-2018.1.382. PMID 30504336
- [Background] Perry DK, Burns JM, Pollinger HS, Amiot BP, Gloor JM, Gores GJ, Stegall MD. Proteasome inhibition causes apoptosis of normal human plasma cells preventing alloantibody production. Am J Transplant. 2009 Jan;9(1):201-9. doi: 10.1111/j.1600-6143.2008.02461.x. Epub 2008 Oct 31. PMID 18976291
- [Background] Palombella VJ, Rando OJ, Goldberg AL, Maniatis T. The ubiquitin-proteasome pathway is required for processing the NF-kappa B1 precursor protein and the activation of NF-kappa B. Cell. 1994 Sep 9;78(5):773-85. doi: 10.1016/s0092-8674(94)90482-0. PMID 8087845
- [Background] Berges C, Haberstock H, Fuchs D, Miltz M, Sadeghi M, Opelz G, Daniel V, Naujokat C. Proteasome inhibition suppresses essential immune functions of human CD4+ T cells. Immunology. 2008 Jun;124(2):234-46. doi: 10.1111/j.1365-2567.2007.02761.x. Epub 2008 Jan 23. PMID 18217957
- [Background] Goldberg AL, Cascio P, Saric T, Rock KL. The importance of the proteasome and subsequent proteolytic steps in the generation of antigenic peptides. Mol Immunol. 2002 Oct;39(3-4):147-64. doi: 10.1016/s0161-5890(02)00098-6. PMID 12200047
- [Background] Ratnasingam S, Walker PA, Tran H, Kaplan ZS, McFadyen JD, Tran H, Teh TC, Fleming S, Catalano JV, Chunilal SD, Johnston A, Opat SS, Shortt J. Bortezomib-based antibody depletion for refractory autoimmune hematological diseases. Blood Adv. 2016 Nov 22;1(1):31-35. doi: 10.1182/bloodadvances.2016001412. eCollection 2016 Nov 29. PMID 29296693
- [Background] Muhsen IN, Alahmari A, Alnahedh M, Alkhudair NA, Samarkandi H, El Fakih R. Bortezomib for immune thrombocytopenia and autoimmune hemolytic anemia. Hematol Oncol Stem Cell Ther. 2020 Dec;13(4):251-254. doi: 10.1016/j.hemonc.2019.05.006. Epub 2019 Jun 10. No abstract available. PMID 31202670
- [Background] Reynaud Q, Durieu I, Dutertre M, Ledochowski S, Durupt S, Michallet AS, Vital-Durand D, Lega JC. Efficacy and safety of rituximab in auto-immune hemolytic anemia: A meta-analysis of 21 studies. Autoimmun Rev. 2015 Apr;14(4):304-13. doi: 10.1016/j.autrev.2014.11.014. Epub 2014 Dec 9. PMID 25497766
- [Background] Danchaivijitr P, Yared J, Rapoport AP. Successful treatment of IgG and complement-mediated autoimmune hemolytic anemia with bortezomib and low-dose cyclophosphamide. Am J Hematol. 2011 Mar;86(3):331-2. doi: 10.1002/ajh.21950. Epub 2011 Jan 26. No abstract available. PMID 21271614
- [Background] Hosoba S, Jaye DL, Cohen C, Roback JD, Waller EK. Successful treatment of severe immune hemolytic anemia after allogeneic stem cell transplantation with bortezomib: report of a case and review of literature. Transfusion. 2015 Feb;55(2):259-64. doi: 10.1111/trf.12815. Epub 2014 Aug 25. PMID 25156334
- [Background] Cao L, Koh LP, Linn YC. Successful treatment of refractory autoimmune hemolytic anemia after allogeneic hematopoietic stem cell transplantation with bortezomib. Leuk Lymphoma. 2018 Oct;59(10):2500-2502. doi: 10.1080/10428194.2017.1421759. Epub 2018 Jan 18. No abstract available. PMID 29345206